CLINICAL TRIAL: NCT06210282
Title: The Effect of Focused Lung Ultrasonography on Antibiotic Prescribing in Patients With Acute Lower Respiratory Tract Infections in Danish General Practice: A Pragmatic Randomised Controlled Trial
Brief Title: The Effect of Focused Lung Ultrasonography on Antibiotic Prescribing in General Practice
Acronym: PLUS-FLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Julie Jepsen Strøm, MD, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N-20230038
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lower Respiratory Tract Infection; Community Acquired Pneumonia
Keywords: Lower Respiratory Tract Infection; Community Acquired Pneumonia; Lung Ultrasound; Point-of-care Ultrasound; General Practice; Antibiotics
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants assigned to the usual care group will receive the general practitoner's usual care of adults (≥ 18 years) presenting with symptoms of an acute lower respiratory tract infection (LRTI) where the GP suspects community-acquired pneumonia. Usual care will be used as a pragmatic comparator to reflect the current standard examinations and care of this patient population in general practices in Denmark. Usual care is recommended to follow applicable guidelines from the Danish Society of General Practitioners and The Doctor's Handbook. Focused lung ultrasound (FLUS) is currently not standard or even a common examination in Danish general practices. Even for GPs already using point-of-care ultrasound on a weekly basis, FLUS is not part of usual care for adults presenting with symptoms of an acute LRTI
  Interventions: Other: Usual Care
- Usual Care + Focused lung ultrasound (FLUS) (Experimental): Participants assigned to the intervention group will receive a focused lung ultrasound examination (FLUS) during the index consultation (day 0) as an addition to usual care.
  Interventions: Diagnostic Test: Focused lung ultrasound (FLUS); Other: Usual Care

INTERVENTIONS:
Diagnostic Test: Focused lung ultrasound (FLUS) — We will use a 14-zone scanning approach. Each hemithorax is divided into anterior, lateral, and posterior surfaces. The anterior and lateral surfaces on each hemithorax are divided into an upper and lower quadrant. The posterior surfaces on each hemithorax are divided into an upper, middle, and lower quadrant. Each quadrant represents a scanning zone. Each scanning zone should be assessed using FLUS. The participating general practitioners use point-of-care ultrasound on a weekly basis before trial commencement and will use the ultrasonography device already available to them.
  Arms: Usual Care + Focused lung ultrasound (FLUS)
Other: Usual Care — Participants assigned to the control group will receive the GP's usual care of adults (≥ 18 years) presenting with symptoms of an acute LRTI where the GP suspects CAP. Usual care will be used as a pragmatic comparator to reflect the current standard examinations and care of these patients in general practices in Denmark. Usual care is recommended to follow applicable guidelines from the Danish Society of General Practitioners (DSAM) and Lægehåndbogen [The Doctor's Handbook].

SUMMARY:
The goal of this randomised controlled trial is to determine if adults presenting with symptoms of an acute lower respiratory tract infection in general practice where the general practitioner suspects CAP, who have FLUS performed as an addition to usual care, have antibiotics prescribed less frequent compared to those given usual care only.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Acute cough (< 21 days).
3. At least one other symptom of acute lower respiratory tract infection (LRTI).
4. The general practitioner suspects a bacterial community-acquired pneumonia.

Exclusion Criteria:

1. Previous antibiotic treatment for the current episode of acute LRTI.
2. The patient is not listed with the general practitioner (no medical record available).
3. The patient is not capable of understanding and signing informed consent.
4. The patient does not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Antibiotics prescribed at index consultation | Day 0
  The primary outcome is the proportion of participants with antibiotics prescribed at index consultation (day 0) reported by the GP at index consultation. We will assess the effect of adding FLUS to usual care on antibiotics prescribed at index consultation by investigating if there is a difference between groups in the proportion of participants with antibiotics prescribed at index consultation..

SECONDARY OUTCOMES:
Daily total LRTI symptom-score | From day 0 until participants have scored 0 in every symptom item, whichever comes first, or up to a maximum of day 21.
  Daily total LRTI symptom-score in groups, calculated as sum of scores of six symptoms (minimum 0 - maximum 36) (mean/median). Participants will be asked to complete a validated LRTI symptom diary every day from day 0 up until day 21. The recorded items include the following six symptoms of LRTI: cough, dyspnea, sputum production, well-being, sleep disturbance, and activity disturbance. The participants will be asked to consider how bad each symptom has been, over the past 24 hours by scoring each symptom on a 7-point Likert-scale (0 = no problem, 1 = very little problem, 2 = slight problem, 3 = moderate problem, 4 = bad problem, 5 = very bad problem, and 6 = as bad as it could be).
Days with symptoms being a "moderate problem" or worse | From day 0 until participants have scored 0 in every symptom item, whichever comes first, or up to a maximum of day 21.
  Number of days with symptoms rated a "moderate problem" or worse by the participants in groups (at least one item with score 3 or above) (mean/median).
Days signed in sick/cancelled work-related activities | From day 0 until the participant has scored 0 in every symptom item, whichever comes first, or up to a maximum of day 21.
  Number of days participants signed in sick/cancelled work-related activities or cancelled leisure activities (mean/median) in groups.
Satisfaction with the index consultation | Day 0
  Proportion of participants satisfied or very satisfied (4 or 5) with the index consultation on a 5-point Likert scale.
Antibiotics prescribed as delayed antibiotic prescription | Day 0
  Proportion of antibiotics prescribed as delayed antibiotic prescriptions at index consultation (day 0).
Antibiotics prescribed during follow-up | Up until day 28
  Proportion of participants with antibiotics prescribed within 7 and 28 days after index consultation.
Re-consultations | Up until day 28.
  Proportion of participants with re-consultations, defined as any primary care contacts (general practice or out-of-hour services), within 28 days after index consultation.
Admission to hospital | Up until day 28.
  Proportion of participants admitted to hospital within 28 days after index consultation.
Complications | Up until day 28.
  Proportion of participants with complications (pleural infection (defined as complicated parapneumonic effusion or empyema), lung abscess, or sepsis) during admission to hospital within 28 days after index consultation.
Other imaging than FLUS performed | Up until day 28.
  Proportion of participants with other imaging than FLUS (any imaging performed in secondary health care services) performed within 28 days after index consultation.
Types of other imaging performed | Up until day 28.
  Types of other imaging than FLUS performed within 28 days after index consultation.
Referred with suspicion of cancer | Up until day 60.
  Proportion of participants referred with suspicion of cancer within 60 days after index consultation.
Diagnoses of cancer | Up until day 60.
  Proportion of participants in groups diagnosed with cancer within 60 days after index consultation.
Spontaneously reported unintended events | Up until day 60.
  Number of spontaneously reported unintended events up until 60 days after index consultation.
Mortality | Up until day 28 and 60.
  All-cause mortality up until day 28 and day 60.

CONTACTS AND LOCATIONS:
Overall Officials: Julie J Strøm, MD, Principal Investigator — Aalborg University
Locations (1):
- Center for General Practice at Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strom JJ, Andersen CA, Bach Jensen M, Laust Thomsen J, Laursen CB, Skaarup SH, Lawaetz Schultz HH, Hansen MP. The effect of focused lung ultrasound on antibiotic prescribing in patients with acute lower respiratory tract infections in Danish general practice (PLUS-FLUS): a pragmatic, randomised controlled, post-market trial. EClinicalMedicine. 2025 Sep 18;88:103518. doi: 10.1016/j.eclinm.2025.103518. eCollection 2025 Oct. PMID 41035797
- [Derived] Strom JJ, Andersen CA, Jensen MB, Thomsen JL, Laursen CB, Skaarup SH, Schultz HHL, Hansen MP. The effect of focused lung ultrasonography on antibiotic prescribing in patients with acute lower respiratory tract infections in Danish general practice: study protocol for a pragmatic randomized controlled trial (PLUS-FLUS). Trials. 2024 May 2;25(1):298. doi: 10.1186/s13063-024-08129-2. PMID 38698471

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06210282/SAP_000.pdf